CLINICAL TRIAL: NCT03811236
Title: Cold-induced Brown Fat Activation and Hepatic Steatosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Florian Kiefer, Associate Professor of Medicine, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1911/2017
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold exposure (Experimental)
  Interventions: Other: Cold exposure
- Room temperature (No Intervention)

INTERVENTIONS:
Other: Cold exposure — Two hours of mild cold exposure using a water-perfused vest
  Arms: Cold exposure

SUMMARY:
In the recent years, research on brown adipose tissue (BAT) revealed that larger amounts as well as higher activity thereof are associated with a favourable metabolic phenotype. Longitudinal studies which applied recurrent cooling sessions demonstrated a high plasticity of BAT which significantly increased in size and activity during these studies. These changes were accompanied by improvements in body fat mass as well as insulin sensitivity. Non-alcoholic fatty liver disease (NAFLD) is estimated to advance to the primary cause of liver cirrhosis and hepatocellular carcinoma in the following years. Besides predisposing genetic and possibly nutritional factors, the insulin resistance syndrome and obesity are the main factors contributing to this excessive hepatic lipid accumulation.

The aim of this study is to investigate whether BAT recruitment via cold-acclimation results in decreased hepatic lipid content in overweight/obese patients with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 28 - 40 kg/m^2
* hepatic lipid content > 10 %

Exclusion Criteria:

* endocrine disease, except treated hypo-/hyperthyroidism and hypertriglyceridemia (<500 mg/dl) and untreated type II diabetes mellitus (fasting glucose < 140 mg/dl)
* use of beta-blockers, alpha-blockers and rilmenidine
* chronic kidney disease
* inflammatory bowel disease
* active malignant disease
* autoimmune disease
* chronic alcohol abuse or alcohol consumption greater than 30g/d for men or 20 g/d for women
* transferrin saturation > 40%
* serum alpha-1 antitrypsin < 90 mg/dl
* serum ceruloplasmin < 20 mg/dl
* positive serology for autoimmune hepatitis
* positive hepatitis serology
* liver cirrhosis
* portal hypertension
* pregnancy
* contraindications for magnetic resonance imaging

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Hepatic lipid content (%) | Six weeks
  Magnetic resonance imaging-proton density fat fraction

SECONDARY OUTCOMES:
Brown adipose tissue volume (ml) / activity (SUVmean) | Six weeks
  18-fluorodeoxyglucose positron emission tomography/ magnetic resonance imaging
Basal metabolic rate (kcal/day/kg fat-free body mass) | Six weeks
  Indirect calorimetry
Cold-induced non-shivering thermogenesis (%) | Six weeks
  Indirect calorimetry: percentage increase in basal metabolic rate before and after cold exposure
Body fat mass (kg) | Six weeks
  Air displacement plethysmography
Insulin sensitivity | Six weeks
  "Matsuda Index" for 2 hour standard oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Florian Kiefer, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No